CLINICAL TRIAL: NCT06314516
Title: Influence of Nutrition and SarcoPenia on Esophageal Cancer ouTcomes (INSPECT Study)
Brief Title: Influence of Nutrition and Sarcopenia on Esophageal Cancer Outcomes
Acronym: INSPECT
Status: Completed | Type: Observational
Sponsor: Benaroya Research Institute (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CRP17122
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer; Sarcopenia
MeSH Terms: conditions — Esophageal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Body Composition: Radiologic assessment of fat and muscle components of body composition at presentation and following initial treatment for esophageal cancer.

SUMMARY:
Prospective multicenter longitudinal (observational) study recruiting from tertiary centers for the surgical management of esophageal cancer; Virginia Mason Medical Center (Seattle, USA) and St Mary's Hospital (Imperial College, London, UK). This is intended to be a pilot study.

DETAILED DESCRIPTION:
Patients undergoing curative treatment for esophageal cancer will be recruited at the time of routine clinical assessment shortly following initial diagnosis and will undergo clinical and radiological evaluation at two study time points: (1) staging investigation (e.g. laparoscopy or endoscopy) and (2) definitive surgical resection. Study time points have been judiciously chosen to coincide with interventions that form part of patient's routine clinical care. It is intended that sampling will occur on the day of each intervention/surgery following a routine period of fasting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following characteristics will be eligible for inclusion in this study:

  * Age 18-90 years
  * Newly diagnosed (prior to treatment) with esophageal and/or gastroesophageal junctional cancer (adeno- or squamous cell carcinoma)
  * Planning to undergo curative treatment, including surgical resection with or without neoadjuvant therapy

Exclusion Criteria:

* Patients with the following characteristics will not be eligible for inclusion in this study:

  * Pregnant females
  * Without malignant esophageal disease
  * Inability or unwillingness to provided informed written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: International cohort of patients presenting with regional {Stage 2 and 3} esophageal cancer who are considered appropriate candidates for surgical therapy.
Sampling Method: Probability Sample
Enrollment: 1717 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Longitudinal variation in body composition | Approximately 1 year
  Establish the effect of patient and disease-specific factors on body composition in a global cohort of patients undergoing esophagectomy for cancer

SECONDARY OUTCOMES:
Patient and disease-specific factors | Approximately 1 year
  Provide a benchmark for future reporting of body composition and to explore the association between body composition and outcomes of esophageal cancer surgery

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Low, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Patient characteristics will be pulled out by three regions, North America, Europe and Asia. Additional anonymized data may be available upon request.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT06314516/Prot_000.pdf
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT06314516/ICF_001.pdf